CLINICAL TRIAL: NCT01666769
Title: Safety and Pharmacokinetics of Micafungin in Children Supported With Extracorporeal Membrane Oxygenation
Brief Title: Pharmacokinetics of Micafungin in Children on Extracorporeal Membrane Oxygenation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kevin Watt (Other)
Responsible Party: Sponsor-Investigator, Kevin Watt, Assistant Professor, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00039552
Record Dates: First submitted 2012-08-14; First posted 2012-08-16 (Estimated); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Invasive Candidiasis
Keywords: Extracorporeal membrane oxygenation; ECMO; Extracorporeal life support; Micafungin; Mycamine; Pharmacokinetics
MeSH Terms: conditions — Candidiasis, Invasive | interventions — Micafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment Dosing (Other): Age group: 0 - <2y, Micafungin 8 mg/kg/day IV
  Interventions: Drug: Micafungin
- Prophylaxis dosing (Other): Age group: 0-<2y, Micafungin 4 mg/kg/day IV
  Interventions: Drug: Micafungin
- Standard of care Dosing (Other): Age group: 2-17.85 y, Micafungin standard of care dosing (decided by treating physician)
  Interventions: Drug: Micafungin

INTERVENTIONS:
Drug: Micafungin — 4 mg/kg/day
  Other Names: Mycamine
  Arms: Prophylaxis dosing
Drug: Micafungin — 8 mg/kg/day
  Other Names: Mycamine
  Arms: Treatment Dosing
Drug: Micafungin — Standard of care Dosing
  Other Names: Mycamine
  Arms: Standard of care Dosing

SUMMARY:
Determine proper dosing of micafungin in children supported with extracorporeal membrane oxygenation (ECMO).

DETAILED DESCRIPTION:
Extracorporeal membrane oxygenation (ECMO) is a cardiopulmonary bypass device that provides life-saving, complete respiratory and cardiac support for children who suffer refractory heart or lung failure. While on ECMO, children are at increased risk of infection, including fungal infection. Antifungal prophylaxis can potentially reduce the burden of disease in children on ECMO. Because fungal infections can result in biofilms that are difficult to treat, treatment includes not only antifungal medications but also removal of any large intravenous lines. However, catheter removal for children on ECMO is impossible; therefore, therapy relies upon optimal antifungal management alone.

Micafungin is an antifungal medication that works well against the most common fungal infections and has been shown to be safe in children. Micafungin may be particularly efficacious in children on ECMO because of the drug's ability to penetrate biofilms. However, the ECMO circuit is known to substantially alter drug levels for many drugs, resulting in important dosing changes. Appropriate micafungin dosing in this setting is unknown and sub-optimal dosing might result in therapeutic and prophylactic failure.

Standard dosing of micafungin are 4 and 2 mg per kilogram of body weight given intravenously once daily for treatment and prophylaxis, respectively. Based on preliminary data and modeling from other studies, investigators hypothesize that 8 and 4 mg per kilogram given once daily will achieve proper drug levels to respectively treat and prevent fungal infections in children under 2 years of age who are supported by ECMO. Because the ECMO circuit should have less of an impact on volume of distribution in larger children, investigators hypothesize that in children from 2 to 18 years old, standard dosing of micafungin will achieve proper drug concentrations.

Investigators hold the FDA investigational new drug application (IND #115255) to give micafungin to children on ECMO at the doses described above. Blood samples will be collected at specific times around the first and fourth micafungin doses to describe the pharmacokinetics and drug extraction by the ECMO circuit.

ELIGIBILITY:
Inclusion Criteria:

* <= 17.85 years at the time of enrollment.
* Sufficient venous access to permit administration of study medication.
* Supported with either venoarterial (VA) or venovenous (VV) ECMO.
* Availability and willingness of the parent/legal guardian to provide written informed consent.
* For treatment dosing arm: confirmed or suspected infection

Exclusion Criteria:

* Subject with a history of anaphylaxis attributed to an echinocandin.
* Any other concomitant condition, which in the opinion of the investigator would preclude a subject's participation in the study.
* Previous participation in this study.
* Pregnancy

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-02-02 (Actual); Study Completion 2016-02-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic primary endpoints | Around the first and fourth doses of micafungin: 0-4h prior to and 0-30 min, 60-90 min, 2-4h, 8-10h, 12-16h, 22-24h after infusion of study drug
  Clearance rate (CL), Volume of distribution (V), Oxygenator extraction efficacy

SECONDARY OUTCOMES:
Safety | From Dose 1 until 7 days after the last dose
  Number of adverse events (any untoward medical occurrence in humans, whether or not considered drug-related, which occurs during the conduct of a clinical trial)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Watt, MD, Principal Investigator — Duke Clinical Research Institute
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States